CLINICAL TRIAL: NCT03408041
Title: Reported Time Between Onset and Diagnosis of Alzheimer's Disease: Correlation With Objective Parameters
Status: Completed | Type: Observational
Sponsor: Murielle Surquin (Other)
Responsible Party: Sponsor-Investigator, Murielle Surquin, Head of clinic, Brugmann University Hospital
Organization: Brugmann University Hospital (Other)
Other Study IDs: CHUB-parameters Alzheimer
Record Dates: First submitted 2018-01-17; First posted 2018-01-23 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer Disease; Objective parameters; Scheltens index
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Alzheimer Disease: Alzheimer Disease patients admitted in the 'Memory Clinic' of the CHU Brugmann Hospital between 01-01-2010 and 31-01-2013. Diagnose according to the Dubois criteria
  Interventions: Other: Medical file data extraction

INTERVENTIONS:
Other: Medical file data extraction — Medical file data extraction

SUMMARY:
The early diagnosis of Alzheimer's disease is essential to enable patients to have access to the available treatments. However, there is a delay between the diagnosis and the onset of symptoms, which can range from 1 year to more than 5 years. In clinical practice, the hippocampal volume, measured by the Scheltens index, is currently used as a marker of the progression of the disease.

The purpose of this study is to determine whether the patient's sex, age and ethnicity can influence the delay in the expression of cognitive troubles reported by the family at the first medical consultation, as well as to determine if there is a correlation between the delay reported by the family and the Scheltens index.

ELIGIBILITY:
Inclusion Criteria:

Alzheimer Disease patients admitted in the 'Memory Clinic' of the CHU Brugmann Hospital between 01-01-2010 and 31-01-2013. Diagnose according to the Dubois criteria

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Alzheimer Disease patients admitted in the 'Memory Clinic' of the CHU Brugmann Hospital between 01-01-2010 and 31-01-2013. Diagnose according to the Dubois criteria
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
Age | Between 01-01-2010 and 31-01-2013
  Age
Sex | Between 01-01-2010 and 31-01-2013
  Sex
Ethnic origin | Between 01-01-2010 and 31-01-2013
  Ethnic origin
Symptoms-diagnose time interval | Between 01-01-2010 and 31-01-2013
  Interval of time between the apparition of the first symptoms, as reported by the family, and the diagnose.
Scheltens scale | Between 01-01-2010 and 31-01-2013
  Evaluation of the hippocampal atrophy by means of magnetic resonance imaging. Scale from 0 (normal) to 4.

CONTACTS AND LOCATIONS:
Overall Officials: Florence Benoit, MD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No